CLINICAL TRIAL: NCT00467454
Title: A Double-Blind, Placebo-Controlled Study of Naltrexone in Pyromania
Brief Title: Naltrexone in the Treatment of Pyromania
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding allocation to different clinical trials.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0703M04084
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Pyromania
Keywords: Pyromania; Fire Setting; Compulsive Fire Setting
MeSH Terms: conditions — Firesetting Behavior | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Naltrexone
  Interventions: Drug: Naltrexone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — daily
  Other Names: Revia
  Arms: 1
Drug: Placebo — daily
  Arms: 2

SUMMARY:
The proposed study will consist of 8 weeks of treatment with either naltrexone or placebo in 10 subjects with pyromania.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the efficacy and safety of naltrexone in pyromania. Ten subjects with DSM-IV pyromania will receive 8 weeks of naltrexone or placebo. The hypothesis to be tested is that naltrexone will be effective in reducing the urges to set fires patients with pyromania. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. men and women age 16-75;
2. current DSM-IV pyromania

Exclusion Criteria:

1. unstable medical illness or clinically significant abnormalities on prestudy laboratory tests or physical examination;
2. history of seizures;
3. myocardial infarction within 6 months;
4. current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
5. clinically significant suicidality;
6. current or recent (past 3 months) DSM-IV substance abuse or dependence;
7. illegal substance within 2 weeks of study initiation;
8. initiation of psychotherapy or behavior therapy from a mental health professional within 3 months prior to study baseline;
9. initiation of a psychotropic medication within 2 months prior to study inclusion;
10. previous treatment with naltrexone; and
11. treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale Modified for Pyromania (P-YBOCS) | At each visit

SECONDARY OUTCOMES:
Pyromania Symptom Assessment Scale (P-SAS); Sheehan Disability Inventory | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States